CLINICAL TRIAL: NCT06047626
Title: Living Well With Lymphoma: Improving Diet Quality to Improve Energy, Sleep and Quality of Life
Brief Title: Living Well With Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: American Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2023.015; HUM00230256 (Other: University of Michigan)
Record Dates: First submitted 2023-04-03; First posted 2023-09-21 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fatigue Reduction Diet- FRD (Experimental): 3 months of individualized counseling of the FRD delivered by registered dietitians, over 8 sessions by phone/video conferencing on fatigue, quality of life, and associated symptoms in persistently fatigued lymphoma cancer survivors
  Interventions: Other: Fatigue Reduction Diet
- General Health Curriculum- GHC (Active Comparator): 3 months of individualized counseling of the attention control (matched for time and frequency of interactions with the FRD) the General Health Curriculum (GHC)
  Interventions: Other: General Health Curriculum

INTERVENTIONS:
Other: Fatigue Reduction Diet — Sessions will be ~15 minutes for 8 sessions. The FRD maintains participants on a diet with their typical caloric intake as assessed at baseline, and replaces some of their calories with the following foods on a daily basis: at least 50% of servings grains to be whole grains (these would replace non-whole grain foods); 5 servings of vegetables (1 leafy green, 1 tomato, and 1 yellow/orange); 2 servings of fruit (1 high in vitamin C), both fruit and vegetables would replace some of the carbohydrates from non-fruit and vegetable sources; 1 serving of fatty fish and or 1 serving of nuts and/or seeds (2 servings of nuts and/or seeds for vegetarians), both the fish, the nuts, and seeds will replace existing sources of fats and proteins in the diet.
  Arms: Fatigue Reduction Diet- FRD
Other: General Health Curriculum — These sessions will be matched counseling method, time spent (~15 minutes per session), for 8 sessions. Registered Dietitians will discuss general health topics with the participant, excluding topics of diet and food.
  Arms: General Health Curriculum- GHC

SUMMARY:
In this study the investigators are proposing to evaluate the efficacy, sustainability, and mechanisms of 3 months of individualized counseling of the FRD delivered by registered dietitians, over 8 sessions by phone/video conferencing on fatigue, quality of life, and associated symptoms in persistently fatigued lymphoma cancer survivors compared to 3 months of individualized counseling of the attention control (matched for time and frequency of interactions with the FRD) the General Health Curriculum (GHC). The investigators will randomize and follow 68 lymphoma cancer survivors; accounting for a ~10% drop out rate to achieve a target of 60 patients that will complete the study. The investigators hypothesize that persistently fatigued lymphoma cancer survivors will experience improvements in fatigue, quality of life, and symptoms commonly associated with fatigue, which are then maintained at 15-months post-enrollment; and decreased CRP and alterations in inflammation-associated DNA methylation consistent with reduced inflammation from following the FRD as compared to the GHC.

DETAILED DESCRIPTION:
26OCT2025- Overall enrollment increased to 100

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18 years and older
* Diagnosis of lymphoma (Hodgkin and non-Hodgkin)
* Have an average persistent fatigue defined as ≥ 4 on the Brief Fatigue Inventory
* Fatigue must be attributed to lymphoma diagnosis
* Fatigue onset must be between 12months before diagnosis and any time after diagnosis
* Fatigue must not be attributed to other disease diagnoses
* Fruit and vegetable intake ≤5.5 servings/day
* Have, or be willing to create, an email address to receive study questionnaires electronically.

Exclusion Criteria:

* Medically unstable
* BMI<18.5 kg/m2
* Have a current untreated diagnosis of mood disorder, e.g., bipolar or major depressive disorder
* Have a current untreated diagnosis of anemia
* Have a current untreated diagnosis of hypothyroidism
* Have an initiation, a cessation or change of treatment of any chronic medications, dietary supplements, behavioral therapy, physical therapy etc., or any planned change of medications, supplements, or therapies during the study
* Have a current diagnoses of cachexia
* Planning on becoming pregnant, currently pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Brief Fatigue Inventory | 3 months after enrollment
  To examine the effect of 3 months of FRD compared to an attention control GHC on persistent fatigue, measured with the Brief Fatigue Inventory. The instrument consists of 9 items, each measuring fatigue on a 0-10 scale, and is calculated from the mean of completed items

SECONDARY OUTCOMES:
Examining the effect of 3 months of FRD compared to an attention control GHC on Quality of life | 3 months after enrollment
  Quality of life, using the Functional Assessment of Chronic Illness Therapy Measurement System, specifically the lymphoma cancer specific instrument. The total score will be our primary outcome. The FACT-G has demonstrated reliability, validity, and responsiveness to change over time.
The effect of 3 months of FRD compared to an attention control GHC on persistent sleep disturbance | 3 months after enrollment
  Using the PROMIS SF v1.0- Sleep Disturb 8b survey
The effect of 3 months of FRD compared to an attention control GHC on persistent pain | 3 months after enrollment
  Using the PROMIS SF v1.1- Pain Interference 8a survey
The effect of 3 months of FRD compared to an attention control GHC on persistent mood | 3 months after enrollment
  Using the PROMIS SF v1.0 Anxiety 7a and Depression 8b surveys
The effect of 3 months of FRD compared to an attention control GHC on persistent sexual function | 3 months after enrollment
  Using the PROMIS Sexual Function Profile v1.0 Mal and Female surveys
Examining the effect of 3 months of FRD compared to an attention control GHC on adherence to program | 3 months after enrollment
  Adherence measured with a food frequency questionnaire (FFQ) and food checklists.
Examining the acceptability of the FRD program- FRD initiation | 3 months after enrollment
  Acceptability via semi-structured interviews (only in the FRD arm), specifically barriers and facilitators to FRD initiation
Number of subjects who withdraw from study (acceptability) | 3 months after enrollment
  Acceptability via withdrawals over the 3-month intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Suzie Zick, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No we would not make individual data just composite data available.